CLINICAL TRIAL: NCT05435495
Title: Mechanisms of Resistance to PSMA Radioligand Therapy: Radiation Resistance Versus Dose
Brief Title: Mechanisms of Resistance to PSMA Radioligand Therapy
Status: Recruiting | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 19553; R01CA235741-03 (NIH)
Record Dates: First submitted 2022-06-22; First posted 2022-06-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: Radioligand Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue and blood samples will be obtained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants undergoing 177Lu-PSMA-617 treatment: Participants undergoing PSMA targeted radioligand therapy with at least four cycles of treatment planned will undergo the following: SPECT/CTs will be performed 24 hours after the first treatment and after the fourth treatment, a tumor biopsy will be performed prior to the first 177Lu-PSMA radioligand therapy, a blood will be drawn prior to treatment for future research, and an optional tumor biopsy and blood draw for future research, may also be obtained at time of progression.
  Interventions: Procedure: Single-photon emission computed tomography; Procedure: Blood Draw; Procedure: Tumor Biopsy

INTERVENTIONS:
Procedure: Single-photon emission computed tomography — Imaging procedure
  Other Names: SPECT/CT
Procedure: Blood Draw — Blood draw for future research tests (45-60 mL).
Procedure: Tumor Biopsy — Guided biopsy of lesion
  Other Names: Biopsy

SUMMARY:
This is a multicenter, correlative study to existing Lutetium based prostate-specific membrane antigen (PSMA)-targeted radioligand therapy (RLT) trials and uses.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the relationship between whole body tumor absorbed dose and response Lutetium based prostate-specific membrane antigen-targeted radioligand therapy (177Lu-PSMA-RLT).

II. To determine the relationship between Post-Operative Radiation Therapy Outcomes Score (PORTOS) score and response to 177Lu-PSMA-RLT.

III. To determine the relative importance of radiation dose (whole body tumor absorbed dose) and radiation sensitivity (PORTOS score) as a marker of response to 177Lu-PSMA-RLT.

EXPLORATORY OBJECTIVES:

I. To develop novel signature of radiation sensitivity.

II. To evaluate tumor biopsies to understand mechanisms of resistance.

III. To understand utility of post-cycle 4 single-photon emission computed tomography (SPECT/CT) to evaluate treatment response.

Study participants will undergo a biopsy and blood draw prior to the initiation of planned therapy, as well as SPECT/CT imaging performed after the first and fourth treatments. One SPECT/CT scan will be performed 24 (+/- 6) after the first treatment, and after the fourth treatment, a 24 +/- 6-hour post-treatment SPECT/CT will be performed. Additionally, study participants may choose to undergo optional biopsy and blood draw at time of progression.

ELIGIBILITY:
Inclusion Criteria:

1. Initiating treatment with Lutetium based PSMA-targeted RLT.
2. Participants must have a PSMA-avid lesion that is accessible to biopsy. Biopsy of newly emerging radiographic metastases is desired and preferable to the biopsy of previously existing lesions whenever possible. Newly emerging lesions are defined as those that are absent on a previous scan, or those demonstrating unequivocal progression since initiation of the last treatment. Biopsies will be performed according to local institutional standards.
3. Patients on warfarin, aspirin, or other anti-coagulants are eligible provided they are deemed able to tolerate discontinuation of anti-coagulation for at least five days prior to the biopsy. Conversion to low molecular weight heparin prior to biopsy is permitted per local standard operating procedures, provided there is approval by the interventional radiologist or the PI.
4. Age >=18 years.
5. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with significant congenital or acquired bleeding disorders (eg von Wildebrand's disease, acquired bleeding factor inhibitors).
2. Patients who are not able to undergo additional study related imaging procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from patients enrolled on Lutetium based PSMA-RLTs and expected to receiving at least four cycles of PSMA-RLT
Sampling Method: Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean whole body tumor absorbed dose (WB Dose) across all metastatic lesions | Up to 6 months
  The unit density sphere model will be implemented using OLINDA, a second-generation personal computer software for internal dose assessment in nuclear medicine to measure mean dose across all metastatic lesions. This approach uses the three time-point SPECT/CTs to create a whole-body dose map, which can then be segmented. Using OLINDA, the total dose to each tumor will be calculated as the integral of activity over time estimated out to 500 hours. Dose will be calculated in gray (Gy).
Median PORTOS score | Up to 6 months
  PORTOS is a gene signature that predicts salvage radiation success. A PORTOS score of zero (called a "low" PORTOS) means it predicts no benefit from salvage radiotherapy. A PORTOS greater than zero (called a "high" PORTOS score) predicts a benefit from salvage radiation.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Memorial Sloan Kettering, New York, New York

IPD SHARING:
Plan to Share IPD: No